CLINICAL TRIAL: NCT03630159
Title: Phase Ib Study of Tisagenlecleucel in Combination With Pembrolizumab in Relapsed/Refractory (r/r) Diffuse Large B-cell Lymphoma (DLBCL) Patients.
Brief Title: Study of Tisagenlecleucel in Combination With Pembrolizumab in r/r Diffuse Large B-cell Lymphoma Patients
Acronym: PORTIA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCTL019J2101; 2018-000973-57 (EudraCT Number)
Record Dates: First submitted 2018-08-01; First posted 2018-08-14 (Actual); Last update posted 2022-08-15 (Actual); Status verified 2022-08

CONDITIONS: Diffuse Large B-cell Lymphoma
Keywords: Lymphoma tisagenlecleucel; Diffuse Large B-cell Lymphoma; CTL019; PORTIA; DLBCL; tisagenlecleucel; pembrolizumab; r/r Diffuse large B-cell Lymphoma; relapsed/refractory Diffuse large B-cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — tisagenlecleucel; pembrolizumab

STUDY DESIGN:
Masking Description: None (Open label)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tisagenlecleucel+Pembrolizumab (Experimental)
  Interventions: Biological: Tisagenlecleucel; Drug: Pembrolizumab

INTERVENTIONS:
Biological: Tisagenlecleucel — Gene modified autologous T cells
  Other Names: CTL019
Drug: Pembrolizumab — anti PD-1

SUMMARY:
A multi-center, open-label, phase Ib study to evaluate the safety and efficacy of the administration of tisagenlecleucel in combination with pembrolizumab in patients with r/r DLBCL who have received 2 or more lines of systemic therapy, including an anti-CD20 and anthracycline based chemotherapy and having failed to or are not candidates for ASCT. The study will consist of 2 parts: dose timing selection part and expansion part.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed DLBCL per local histopathology assessment.
* Relapsed or refractory disease after having recieved 2 or more lines of systemic therapy, including anti-CD20 and anthracycline based chemotherapy, and either having progressed after (or relapsed after) ASCT, or being not candidates for or not consenting to ASCT.
* Measurable disease at time of enrollment
* ECOG performance status that is either 0 or 1 at screening.

Exclusion Criteria:

* Patients with Richter's transformation, and Burkitt lymphoma, and primary DLBCL of CNS.
* Prior treatment with any prior anti-CD19/anti-CD3 therapy, or any other anti-CD19 therapy.
* Patients with active CNS involvement are excluded, except if the CNS involvement has been effectively treated and provided that local treatment was >4 weeks before enrollment.
* Prior allogeneic HSCT.
* Unstable angina and/or myocardial infarction and/or coronary artery bypass graft (CABG), or stroke within 6 months prior to screening, and/or impaired cardiac function or clinically significant cardiac disease
* Patients with a history of prior treatment with anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4 antibodies, other immune checkpoint inhibitors.
* History of interstitial lung disease or (non-infectious) pneumonitis that required oral or intravenous steroids (other than COPD exacerbation) or current pneumonitis.

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-10-09 (Actual); Primary Completion 2021-07-20 (Actual); Study Completion 2021-07-20 (Actual)

PRIMARY OUTCOMES:
Percent of participants recieving pembrolizumab per protocol schedule | 21 days after first pembrolizumab infusion
Dose Timing part: Incidence of dose limiting toxicities (DLTs) | 21 days after first pembrolizumab infusion
Expansion part: Overall response rate (ORR) | 3 month post tisagenlecleucel infusion

SECONDARY OUTCOMES:
Duration of Response (DOR) | 24 months
Progression Free Survival (PFS) | 24 months
Overall Survival (OS) | 24 months
In vivo cellular kinetics of tisagenlecleucel in blood, bone marrow, lymph nodes and other tissues by qPCR and flow cytometry | 24 months
Impact of pembrolizumab dosing strategy on the cellular kinetics of tisagenlecleucel by qPCR and flow cytometry | 24 months
Immunogenicity measured by antibody titres specific to tisagenlecleucel molecule and by the presence of T lymphocytes activated by the tisagenlecleucel protein | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (5):
- United States (3):
  - Emory University School of Medicine SC CTL019, Atlanta, Georgia
  - University of Chicago Medical Center Hematology and Oncology, Chicago, Illinois
  - University of Kansas Hospital and Medical Center U of Kansas Cancer Center, Kansas City, Kansas
- Novartis Investigative Site, Vienna, Austria
- Novartis Investigative Site, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jaeger U, Worel N, McGuirk JP, Riedell PA, Fleury I, Du Y, Han X, Pearson D, Redondo S, Waller EK. Safety and efficacy of tisagenlecleucel plus pembrolizumab in patients with r/r DLBCL: phase 1b PORTIA study results. Blood Adv. 2023 Jun 13;7(11):2283-2286. doi: 10.1182/bloodadvances.2022007779. PMID 36044388
- [Derived] Ernst M, Oeser A, Besiroglu B, Caro-Valenzuela J, Abd El Aziz M, Monsef I, Borchmann P, Estcourt LJ, Skoetz N, Goldkuhle M. Chimeric antigen receptor (CAR) T-cell therapy for people with relapsed or refractory diffuse large B-cell lymphoma. Cochrane Database Syst Rev. 2021 Sep 13;9(9):CD013365. doi: 10.1002/14651858.CD013365.pub2. PMID 34515338
- See also: Novartis results database — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17956
- See also: A Plain Language Trial Summary is available on novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=1106